CLINICAL TRIAL: NCT05097144
Title: Performance of Two Toric Silicone Hydrogel Contact Lenses
Brief Title: Performance of Toric Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-128
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Results first posted 2022-08-24 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2022-10

CONDITIONS: Astigmatism; Myopia
MeSH Terms: conditions — Astigmatism; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, then Lens B (Experimental): Participants wore Lens A for one month and then wore Lens B for one month.
  Interventions: Device: Lens A (fanfilcon A); Device: Lens B (asmofilcon A)
- Lens B, then Lens A (Experimental): Participants wore Lens B for one month and then wore Lens A for one month.
  Interventions: Device: Lens A (fanfilcon A); Device: Lens B (asmofilcon A)

INTERVENTIONS:
Device: Lens A (fanfilcon A) — Daily wear for one month
Device: Lens B (asmofilcon A) — Daily wear for one month

SUMMARY:
The purpose of this study was to evaluate the clinical performance and subjective lens handling (insertion and removal) of two toric silicone hydrogel contact lenses after one month of daily wear each.

DETAILED DESCRIPTION:
This was a prospective, randomized, double masked, bilateral, crossover study. Participants were expected to attend 6 scheduled visits over a period of approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Is not a habitual wearer of either study lens
* Has a contact lens spherical prescription between +4.00 to - 10.00 (inclusive). Best corrected visual acuity of 20/30 or better in either eye
* Have contact lens prescription of no less than -0.75D of astigmatism and no more than -2.25 D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

A person will be excluded from the study if he/she:

* A person was excluded from the study if he/she:
* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -2.50 D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:
* Pathological dry eye or associated findings
* Pterygium, pinguecula, or corneal scars within the visual axis
* Neovascularization > 0.75 mm in from of the limbus
* Giant papillary conjunctivitis (GCP) worse than grade 1
* Anterior uveitis or iritis (past or present)
* Seborrheic eczema, Seborrheic conjunctivitis
* History of corneal ulcers or fungal infections
* Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Velázquez Guerrero, MSc, FIACLE, Principal Investigator — National Autonomous University (UNAM)
Locations (1):
- National Autonomous University (UNAM), Mexico City, Código, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single investigative site located in Mexico City, Mexico.
Groups:
- Lens A, Then Lens B: Participants first wore Lens A for one month and then wore Lens B for one month.
- Lens B, Then Lens A: Participants first wore Lens B for one month and then wore Lens A for one month.
Period: Period 1 (One Month)
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Period 2 (One Month)
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all study participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling (Insertion and Removal)
Description: Subjective lens handling measured ease of insertion and removal on a scale of 0-10, where 10=better performance.
Time Frame: 1 month
Population: All participants who were exposed to study lenses and completed each study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Participants that received Lens A during either the first or second period of the study.
- Lens B: Participants that received Lens B during either the first or second period of the study.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 36 | 36
units on a scale | 9.47 (1.00) | 8.33 (1.54)

ADVERSE EVENTS:
Time Frame: For the duration of the study, approximately two months.
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT05097144/Prot_SAP_000.pdf